CLINICAL TRIAL: NCT02119390
Title: Targeting Enhanced Adherence to Medication: A Pilot Study in Adolescents and Young Adults With Human Immunodeficiency Virus (HIV)
Brief Title: Medication Adherence in Human Immunodeficiency Virus (HIV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P1TEAM
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: adolescents; young adults; medication adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Other): Participants in the Standard Care group will complete a demographic questionnaire at the time of consent as well as other questionnaires during the course of the study. They will receive standard clinical care.
  Interventions: Other: Demographic Questionnaire; Other: Questionnaires
- Pill Trial+ (Experimental): Participants in the Pill Trial+ group will complete a demographic questionnaire at the time of consent as well as other questionnaires during the course of the study. They will receive standard clinical care plus three 25-minute individualized, behavioral, staff-delivered intervention sessions at HAART initiation, and 1-, and 3-month follow-up visits. Two brief booster sessions will also be provided following sessions 1 (in clinic) and 2 (by phone).
  Interventions: Behavioral: Staff-delivered intervention sessions; Other: Demographic Questionnaire; Other: Questionnaires

INTERVENTIONS:
Behavioral: Staff-delivered intervention sessions — In addition to standard clinical care, participants in the Pill Trial+ arm will receive staff-delivered intervention sessions individualized for each participant at HAART initiation, 1-month, and 3-month follow-up. Two booster sessions will also be provided at two weeks following intervention session 1 (in clinic) and intervention session 2 (by phone) to assess any difficulties using the created adherence plans.
  Arms: Pill Trial+
Other: Demographic Questionnaire — Participants will complete a questionnaire developed for the purposes of the current study assessing basic background information.
Other: Questionnaires — Self-reported adherence, health-related quality of life and other questionnaire measures will be administered using a password protected laptop the same day as participants' regularly scheduled outpatient clinic appointments.

SUMMARY:
Although effective treatments are currently available to treat human immunodeficiency virus (HIV), the retrovirus leading to acquired immune deficiency syndrome (AIDS), strict adherence to the treatment regimen is required. Nonadherence to highly active antiretroviral therapy (HAART) regimens is well documented in individuals with HIV. This is especially true for adolescents and young adults (AYA), where rates of adherence range from 20 to 100%. Nonadherence has significant implications for subsequent treatment response and health outcomes, including poor virologic response, development of drug resistance, and mortality. Of note, previous research has suggested that every 1% increase in nonadherence is related to a 2% increased likelihood of detectable viral load (VL) in youth with behaviorally acquired HIV. Furthermore, higher VL is the most salient variable related to increased risk of virus transmission. Thus, nonadherence to HAART is a significant public health issue.

The objective of the proposed research plan is to systematically examine an individualized, behavioral intervention targeting HAART nonadherence in AYAs initiating HAART. The current intervention will support AYA participation in brief, staff-delivered instruction in adherence-promotion skills. Individualized behavioral analysis and motivational interviewing will be applied to provide effective solutions for current barriers to HAART adherence before and after HAART initiation, as recommended by the Panel on Antiretroviral Guidelines for Adults and Adolescents.

DETAILED DESCRIPTION:
The proposed pilot study will utilize a randomized controlled trial to estimate the feasibility, acceptability, and preliminary efficacy of a novel intervention for AYAs diagnosed with behaviorally-acquired HIV initiating HAART.

Standard care for HIV at St. Jude Children's Research Hospital (SJCRH) includes a placebo pill trial to assess patient readiness for therapy prior to starting HAART. Participants on this study will be randomized to either: a control arm of standard therapy, or standard therapy plus an individualized behavioral, staff-delivered intervention (Pill Trial+).

Participants in the control arm will receive standard clinical care. Participants in the Pill Trial+ arm will receive standard therapy plus three 25-minute individualized, behavioral, staff-delivered intervention sessions at HAART initiation, and 1-, and 3-month follow-up visits. Two brief booster sessions will also be provided to the Pill Trial+ arm following sessions 1 (in clinic) and 2 (by phone). In-person intervention sessions and all questionnaires will be completed in conjunction with scheduled clinical care visits. Sessions and measures will be completed by phone at designated time points if a participant becomes unavailable to return to clinic due to extenuating circumstances.

As recommended by Panel guidelines, discussion of placebo pill trial adherence during the first 25-minute session will provide a novel mechanism to discuss barriers to adherence and provide intervention prior to HAART initiation. Remaining sessions will promote adherence following HAART initiation using behavioral problem-solving and motivational interviewing strategies.

Primary Objective:

* To estimate a) rate of consent to the randomized trial and b) differences between the intervention and control conditions with respect to HAART adherence, as measured by pill count.

Secondary Objectives:

* To estimate differences between the intervention and control conditions with respect to other measures of adherence, including HAART self-reported adherence, HAART pharmacy refill, and clinic attendance.
* To examine disease and patient-reported outcomes during the first 6 months following HAART initiation and their relationship to participation in the Pill Trial+ intervention.

ELIGIBILITY:
Inclusion Criteria:

* Behaviorally acquired HIV diagnosis, confirmed via medical chart review.
* Currently followed in the St. Jude Children's Research Hospital (SJCRH) HIV clinic.
* Initiating HAART.
* Recommended a placebo trial.
* 13-24 years of age at time of study entry.
* If 15 years of age or over, willing to give informed consent. If under the age of 15, willing to give assent and accompanied by legal guardian/representative to give informed consent.
* Fluent in English

Exclusion Criteria:

* Previous HAART exposure.
* Unable to understand English and/or not cognitively intact (known IQ < 70) such that the study questionnaires cannot be understood and completed.
* Pregnant female.
* Enrolled on another protocol that excludes participation in this study.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Rate of consent to trial participation | Day 1
Pill count values compared between arms | 3 months post-HAART initiation
  Using Fisher Exact tests
Pill count values compared between arms | 6 months post-HAART initiation
  Using Fisher Exact tests

SECONDARY OUTCOMES:
Adherence rates compared between groups | 3 months post-HAART initiation
  Self-reported adherence rates, pharmacy refill, and clinic attendance will be included in this analysis. Fisher exact tests will be performed to compare adherence rates between groups.
Patient outcome | 6 months following HAART initiation
  Disease and patient-reported outcomes will be examined as well as their relationship to participation in the Pill Trial+ intervention. Viral load (VL), CD4 count/%, health-related quality of life (HRQOL) scores, and beliefs about medication (BAM) scores will be analyzed. Mixed effects models will be employed to explore the efficacy of the intervention on virologic response, HRQOL, and medical beliefs. VL, CD4 count/%, HRQOL, and beliefs will be used as the response variables, respectively, while time since treatment, intervention, and their interaction will be included as covariates.
Adherence rates compared between groups | 6 months post-HAART initiation
  Self-reported adherence rates, pharmacy refill, and clinic attendance will be included in this analysis. Fisher exact tests will be performed to compare adherence rates between groups.
Change in adherence rates compared between groups | Baseline through 6 months post-HAART initiation
  Self-reported adherence rates, pharmacy refill, and clinic attendance will be included in this analysis. Mixed effects models and logistic link will be used to examine differences between groups adherence data and within-subject changes in adherence over time.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Wilkins, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Ingerski LM, Means B, Wang F, Zhang H, Patel N, Gaur AH, Wilkins ML. Preventing Medication Nonadherence of Youth (13-24 Years) With HIV Initiating Antiretroviral Therapy. J Adolesc Health. 2021 Oct;69(4):644-652. doi: 10.1016/j.jadohealth.2021.04.006. Epub 2021 May 28. PMID 34059425
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols